CLINICAL TRIAL: NCT05401240
Title: Cardiopulmonary Exercise Test as an Incentive to Outpatient Cardiac Rehabilitation for Acute Coronary Syndrome Survivors
Brief Title: Using Cardiopulmonary Exercise Test as an Incentive to Outpatient Cardiac Rehabilitation for Acute Coronary Syndrome Survivors.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE22225A
Record Dates: First submitted 2022-05-29; First posted 2022-06-02 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Acute Coronary Syndrome
Keywords: cardiac rehabilitation; cardiopulmonary exercise testing
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CEPT informed (Experimental): the patient is informed and asked to returned to the outpatient department (OPD) in order to received cardiac rehabilitation, as well as to take an important examination (cardiopulmonary exercise testing) for his/her cardiorespiratory fitness.
  Interventions: Behavioral: information reveal
- CPET not informed (No Intervention): the patient is asked to returned to the outpatient department (OPD) in order to received cardiac rehabilitation, but not informed about the cardiopulmonary exercise testing.

INTERVENTIONS:
Behavioral: information reveal — the experimental group will be informed that there will be an important examination about his/her cardiopulmonary fitness condition at the outpatient department (OPD)
  Arms: CEPT informed

SUMMARY:
Exercise-based cardiac rehabilitation is a class I recommendation for acute coronary syndrome (ACS) patients. However, participate rate of outpatient rehabilitation is quite low and remains a global issue. The study is to propose a strategy in order to encourage post-ACS patients to participate in the outpatient cardiac rehabilitation.

DETAILED DESCRIPTION:
Background: exercise-based cardiac rehabilitation is a class I recommendation for acute coronary syndrome (ACS) patients. However, participate rate of outpatient rehabilitation is quite low and remains a global issue. The study is to propose a strategy in order to encourage post-ACS patients to participate in the outpatient cardiac rehabilitation.

Hypothesis: cardiopulmonary exercise test (CPET) incentives ACS survivors to participate in outpatient cardiac rehabilitation.

Objectives: 200 ACS survivors who are eligible for cardiac rehabilitation will be allocated randomly into control and experimental groups.

Method: before discharge, both control and experimental groups will be informed of the importance of cardiac rehabilitation and invited to participate the outpatient rehabilitation. The experimental group will also be told that an important examination, i.e. the CPET, will be performed in order to evaluate their heart function at the outpatient department (OPD).

Primary outcome: the presence of ACS survivors at the OPD of rehabilitation in order to receive the rehabilitation/CPET.

Secondary outcomes: the adherence to cardiac rehabilitation, defined as completing a full course of cardiac rehabilitation (6 sessions) or home-based exercise.

Factors that might influence the presence of ACS survivors at OPD of rehabilitation will also be recorded and analyzed, including:

* Patient characteristics: age, sex, body mass index (BMI), cardiovascular disease (CVD) risk factors
* Electrocardiography (ECG): ST elevation myocardial infarction (STEMI) or non ST elevation myocardial infarction (NSTEMI)
* Lab data: peak troponin level.
* Days of hospitalization. Statistics: t-test, ANOVA

ELIGIBILITY:
Inclusion Criteria:

* acute coronary patients

Exclusion Criteria:

* acute illness that stayed in hospital for more than 2 weeks.
* patients who received surgical intervention
* severe complications (ex. respiratory failure, stroke, acute renal failure)
* contraindications of cardiopulmonary exercise testing
* patients who cannot perform the cardiopulmonary exercise testing

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
the return rate | scheduled appointment time, about 2 to 4 weeks after discharge
  patient that did return to the OPD for examination and cardiac rehabilitation

SECONDARY OUTCOMES:
the adherence | 6 months after discharge
  the percentage of patients that keep taking cardiac rehabilitation for more than one session

CONTACTS AND LOCATIONS:
Overall Officials: Yuchun Lee, MD, Study Director — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No